CLINICAL TRIAL: NCT05350397
Title: How Important Is Acupressure Application in Balancing Heart Rate and Blood Pressure in the Treatment of Atrial Fibrillation? Single-Blind Randomized Experimental Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, AYSE SOYLU, Principal Investigator, Kahramanmaras Sutcu Imam University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KSUanestezia
Record Dates: First submitted 2022-04-06; First posted 2022-04-28 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Atrial Fibrillation
Keywords: Acupressure; atrial fibrillation; blood pressure; heart rate; randomized controlled trial; nursing care
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: Groups with the same trait random, independent, random, application and separated as the control group. Intervention is applied to a group, others are not interfered with, the results are followed by are compared.
  It was performed as a single-blind, pretest-posttest placebo, randomized, parallel-controlled experimental study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Acupressure group (Experimental): The patients in the intervention group were informed about what acupressure was and why it was applied. An acupressure wristband was correctly worn on both wrists to provide patients with adequate pressure on the HT7 point for 5 minutes
  Interventions: Other: How Important Is Acupress Applyıng In Atrıal Fıbrılatıon Treatment?
- Placebo Group (Placebo Comparator): Patients in the placebo group were informed about what acupressure was and why it was applied. In order not to apply pressure to the Shenmen (HT7) pressure point in the patients in this group, the acupressure wristband was placed on both wrists in an inverted and loose manner and the wristband was worn for 5 minutes, the procedure was completed.
  Interventions: Other: How Important Is Acupress Applyıng In Atrıal Fıbrılatıon Treatment?
- Control group (No Intervention): No procedure was applied to the patients in the control group. The patients received routine treatment and care.

INTERVENTIONS:
Other: How Important Is Acupress Applyıng In Atrıal Fıbrılatıon Treatment? — The acupressure wristband was correctly attached to the Experimental Group and acupressure was applied. The placebo group was fitted with an inverted and loose acupressure wristband. No intervention was applied to the control group.
  Arms: Acupressure group; Placebo Group

SUMMARY:
Atrial fibrillation is a common cardiac arrhythmia affecting 1-2% of the population. This rate is expected to increase in the next 30 years. The aim of this study is to determine the effect of acupressure applied to patients with chronic atrial fibrillation on blood pressure and heart rate.

This study was designed as a randomized, placebo-controlled experimental study. As a result of the power analysis, 3 groups were formed, each consisting of 23 subjects. No procedure was applied to the control group before and after the measurements. In patients in the placebo group, an inverted and loose acupressure wristband was attached to the Shenman point to avoid applying pressure to any part of the wrist. Acupressure wristbands were applied towards the Shenmen point to provide adequate pressure to the patients in the intervention group and acupressure was applied twice a day. Acupressure was applied 4 times in two days.

DETAILED DESCRIPTION:
1. INTRODUCTION Atrial fibrillation (AF) is a commonly encountered cardiac arrhythmia, which affects 1-2% of the population and this rate is expected to increase within the next 30 years. The Framingham study, which was started in 1949 and is still ongoing, supports this predicted increase by stating that prevalence will increase together with age. In developing countries, the mean age of patients with AF is increasing, and is currently reported as in the range of 75-85 years . AF is seen in males two-fold more than in females . Causing stroke or long-term symptoms such as chest pain, shortness of breath, palpitations, listlessness, fatigue, insomnia and activity intolerance, AF reduces quality of life .

   There are 3 basic goals in AF treatment. These are control of heart rate, prevention of the risk of emboli and the treatment of arrhythmia. AF treatment should be reliable and low cost, and previous studies have shown supportive treatments which are low-cost, easy to apply, and have no side-effects. In particular, there are studies showing that acupuncture is effective in providing heart rate and arrhythmia control in AF. Acupressure, which is defined as non-invasive acupuncture is a treatment method that is applied using an acustimulation device or by applying physical pressure on certain points of the body with the fingers, hand, palm of the hand, wrist, or with a wristband, to regulate the disrupted energy balance through the energy channels of the body. Although it shows all the effects of acupuncture, it is less known than acupuncture, if it is not applied in accordance with the guideline guidelines, it may cause undesirable situations.

   It has been emphasised in literature that by stimulating acetylcholine, dopamine and encephalon expression, acupressure is effective in muscle relaxation and regulating blood circulation. It has been reported that the application of acupressure to patients has reduced back pain and headache, pain related to osteoarthritis, musculoskeletal system pain, neck pain, and pre and postoperative pain, and because of the reflexive effect of acupressure, has reduced nausea and vomiting by increasing the efficacy of the hypothalamus, which is an extrapyramidal pathway, has balanced the heart rate and reduced sleep disorders.

   As acupressure is not invasive, the acupressure training received within the scope of nursing care can be comfortably applied . However, there have been few studies of nurses on this subject, and there is a need for studies with a high level of evidence.

   Aim The aim of this study was to determine the effect on blood pressure and heart rate of acupressure applied to the Shenman (HT7) point in individuals with chronic AF.

   1.1 Research hypotheses H01: Acupressure applied to the Shenmen (HT7) acupuncture point would have no effect on systolic blood pressure in individuals with AF.

   H02: Acupressure applied to the Shenmen (HT7) acupuncture point would have no effect on diastolic blood pressure in individuals with AF.

   H03: Acupressure applied to the Shenmen (HT7) acupuncture point would have no effect on reducing heart rate in individuals with AF.

   H11: Acupressure applied to the Shenmen (HT7) acupoint has an effect on systolic blood pressure in individuals with AF.

   H12: Acupressure applied to the Shenmen (HT7) acupoint has an effect on diastolic blood pressure in individuals with AF.

   H13: Acupressure applied to the Shenmen (HT7) acupuncture point is effective in reducing heart rate in individuals with AF.
2. METHOD

2.1. Study Design and Patient Selection This study was carried out as a pretest-posttest placebo, randomized, parallel controlled experimental study conducted between 20.02.2018 and 20.07.2018 in Kahramanmaraş Sütçü İmam University Health Practice and Research Hospital Cardiology Intensive Care Unit. In the cardiology department, there are 3 intensive care units, 4 isolation rooms, a total of 27 patient beds. Provides tertiary treatment and care services.

In order to specialize in Acupressure, the researcher attended the acupressure course organized by the Antalya Health and Nature Therapies Association on February 9-10, 2018, which included 16 hours of theoretical and practical courses, and received the acupressure certificate. The researcher also attended an 8-hour basic electrocardiography (ECG) course and received an EKG course participation certificate.

Inclusion criteria were patients with chronic AF, >18 years of age, fully conscious, oriented and cooperative, with a heart rate of 70-120 beats/min, and no history of recent open heart surgery.

Patients with renal failure (which causes deterioration of heart rhythm and structure), liver failure (which affects hemodynamic balance) or hyperthyroidism (increased pulse rate) were excluded from the study.

2.2. Sample selection Between 20.02.2018 and 20.07.2018, a total of 81 patients were treated in the ICU, and 12 of them were excluded from the study because they did not meet the inclusion criteria. Thus, 69 patients were included in the study . Power analysis was performed using G Power 3.1 software to determine the number of patients to be included in the placebo, intervention, and control groups. The analysis showed 69 patients in each group with 23, d:1.3344, an α-type error estimate of 0.05, and a power of 100% .

2.3. Randomization and Blinding There were three cardiology intensive care units in the hospital where the research was conducted. We recruited placebo, control and experimental groups from different intensive care units so that the patients were not affected by each other. In this case, each group had to be in the same intensive care unit. We used a system to select which ICUs would be placebo, control, or experimental to ensure randomisation. We write the numbers 1, 2 and 3 on a piece of paper and put them in a bag. The groups were removed from the bag by an impartial nurse working in the ICU (Akbarnezhad et al., 2019). Then, we divided the patients into groups from a random number table according to the order of hospitalization until the sample power was obtained. The identities of the patients participating in the study were kept confidential. In conclusion, this study was conducted as a pretest-posttest placebo, randomized, parallel controlled experimental study.

2.4. Data collection tools In this study, data were collected using the patient information form and data registration form.

2.4.1. Patient Information Form It includes information such as age, height, weight, education level, marital status, occupation, employment status, other people they live with, medications they use, and social security status of the patients included in the study.

2.4.2. Data Registration Form It is a form developed by researchers to record blood pressure and pulse values before and after the procedure.

2.5. Process and Interventions

2.5.1. Placebo Group Patients in the placebo group were informed about what acupressure was and why it was administered, and were told that they were in a study examining the effect of acupressure on blood pressure and heart rate. In this group, the acupressure wristband was placed on both wrists upside down and loosely in order not to apply pressure to the Shenmen (HT7) pressure point, and the wristband was worn for 5 minutes, and the procedure was completed . Blood pressure and heart rate values were recorded from the monitor before and after wearing the wristband at 09:00 in the morning and at 15:00 in the afternoon for two consecutive days .

2.5.2. Acupressure Group Patients in the intervention group were informed about what acupressure was and why it was applied, and were told that they were in a study examining the effect of acupressure on blood pressure and heart rate. An acupressure wristband was correctly fitted on both wrists to provide adequate pressure to the HT7 point for 5 minutes . Blood pressure and heart rate values were recorded from the monitor before and after the acupressure application at 09:00 in the morning and at 15:00 in the afternoon with a wristband for two consecutive days. All data measured in this study were collected from the devices and no manual measurements were made.

2.5.3. Control Group No procedure was applied to the patients in the control group. The patients in the control group, on the other hand, were told that only blood pressure and pulse values would be measured without giving any information about acupressure within the scope of the study . The patients received routine treatment and care.

2.6. Security assessment Before, during and after the acupressure application, the pulse and blood pressure of the patients were continuously monitored in terms of the possibility of acupressure application to the heart point to have a negative effect on the pulse and blood pressure. During the application of acupressure, the patients were followed up for signs such as bradycardia, hypotension, and discomfort. Since the acupressure wristband may impair circulation in the arm, the patients were checked for side effects such as cyanosis, hematoma, and wrist pain. No complications developed in any patient.

Acupressure was applied to the patients 4 times in total at 09:00 and 15:00 on the 1st and 2nd days. Blood pressure and heart rate were measured 8 times before and after each procedure.

2.6.1. Acupressure Practice Guide Acupressure application guide was created as a result of expert opinion and literature review.

* The patients were informed that acupressure would be applied twice, at 09:00 and 15:00 on the same day.
* Care was taken to ensure that there was an interval of 6 hours between acupuncture applications.
* Acupressure was applied 4 times in total at 09:00 and 15:00 on two consecutive days.
* The patients were told that they may feel slight pain and pressure when pressure is applied with the acupressure wristband, and that the procedure can be terminated at any time if they feel uncomfortable.
* Acupuncture points were determined in each patient using their own fingers.
* In order not to make the application on a full stomach, it was applied before the meals or at least 1 hour after the meal.
* Care was taken to ensure that the application area was suitably lit, quiet and adequately ventilated.
* Care was taken to ensure that the application area was clean and dry.
* Patient privacy was respected.
* The patients were placed in the supine position during the application.
* Before the application, 1-2 minutes of relaxation massage (effusion) was applied to the acupressure areas.
* Following the relaxation massage, an acupressure wristband was applied to the HT7 point, the chronometer was started, and the acupressure wristband was removed after 5 minutes.
* After the procedure, the patients were placed in the semi-Fowler position.

2.7. Ethical Approval Approval for the study was obtained from Kahramanmaraş Sütçü İmam University Faculty of Medicine Clinical Research Ethics Committee (decision dated 31.01.2018 and numbered 18). On February 20, 2018, the necessary permission for the research was obtained from the rector of the same university. Informed consent was obtained from all participants participating in the study.

2.8. Statistical analysis The data obtained in the study were statistically analyzed using the Statistical Package for Social Sciences (SPSS) vn. 25.0 software. Descriptive statistics were expressed as mean ± standard deviation (SD), number (n) and percent (%). Kruskal Wallis Analysis of Variance, Fisher Chi-square test, Posthoc and Wilcoxon tests were used in the evaluations. The results were stated at the 95% confidence interval. A p value of <0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion criteria were patients with chronic AF

* >18 years of age
* Fully conscious
* Oriented and cooperative
* Heart rate of 70-120 beats/min
* No history of recent open heart surgery

Exclusion Criteria:

* Patients with renal failure (which causes deterioration of heart rhythm and structure)
* Liver failure (which affects hemodynamic balance)
* Hyperthyroidism (increased pulse rate) were excluded from the study

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2018-02-20 (Actual); Primary Completion 2018-02-20 (Actual); Study Completion 2018-07-20 (Actual)

PRIMARY OUTCOMES:
Investigation of the effect of acupressure applied to patients with Atrial Fibrillation on systole blood pressure, diastolic blood pressure and heart rate | 6 months
  The first criterion was planned to examine and report the effect of acupressure on systole blood pressure.

SECONDARY OUTCOMES:
Investigation of the effect of acupressure applied to patients with Atrial Fibrillation on systole blood pressure, diastolic blood pressure and heart rate | 6 months
  The first criterion was planned to examine and report the effect of acupressure on diastole blood pressure.

OTHER OUTCOMES:
Investigation of the effect of acupressure applied to patients with Atrial Fibrillation on systole blood pressure, diastolic blood pressure and heart rate | 6 months
  The first criterion was planned to examine and report the effect of acupressure on heart rate.

CONTACTS AND LOCATIONS:
Locations (1):
- KahramanmarasSIU, Kahramanmaraş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- Available data/document: REFERENCE: REFERENCE — https://pubmed.ncbi.nlm.nih.gov/30982782/
- Available data/document: REFERENCE: REFERENCE — http://www.journalagent.com/tkd/pdfs/TKDA_35_70_76_127.pdf
- Available data/document: REFERENCE: REFERENCE — http://pubmed.ncbi.nlm.nih.gov/30982782/
- Available data/document: REFERENCE: REFERENCE — http://dergipark.org.tr/tr/pub/ikcusbfd/issue/60165/705219
- Available data/document: REFERENCE: REFERENCE — http://www.journalagent.com/tkd/pdfs/TKDA_37_60_1_10.pdf
- Available data/document: REFERENCE: REFERENCE — http://pubmed.ncbi.nlm.nih.gov/18992625/
- Available data/document: REFERENCE: REFERENCE — http://www.ncbi.nlm.nih.gov/books/NBK72567/
- Available data/document: REFERENCE: REFERENCE — http://doi.org/10.1016/j.ctcp.2021.101304
- Available data/document: REFERENCE: REFERENCE — http://doi.org/10.1097/HNP.0000000000000384
- Available data/document: REFERENCE: REFERENCE — http://pubmed.ncbi.nlm.nih.gov/23981400/